CLINICAL TRIAL: NCT02787564
Title: Studie Zum Einfluss Der Bereitstellung Von Kostenlosem Favorisiertem Obst Und Gemüse Auf Das Ernährungsverhalten
Brief Title: Offering Free Fruits and Vegetables to Men at Risk of Poverty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Principal Investigator, Nanette Stroebele-Benschop, Professor, University of Hohenheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: free F+V
Record Dates: First submitted 2016-05-25; First posted 2016-06-01 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Dietary Habits
Keywords: fruit, vegetables
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Free Fruit and Vegetables (Experimental): After baseline assessment of food intake patterns, the intervention will consist of providing free fruits and vegetables of their choice for a period of four weeks which will be provided fresh each week. At baseline and at the end of the 4-week period, a FFQ, two 24h-recalls and a questionnaire on consumed fruit and vegetable variety will be administered.
  Interventions: Behavioral: Intervention Group
- Control Goup (No Intervention): At baseline and at the end of the 4-week period, a FFQ, four 24h-recalls and a questionnaire on consumed fruit and vegetable variety will be administered. At the end of the intervention period they receive once a basket of free fruits and vegetables.

INTERVENTIONS:
Behavioral: Intervention Group — The intervention consists of providing free fruits and vegetables of the participants' liking for a period of 4 weeks. Each week, a total of 2 portions of either fruits and/or vegetables per day will be provided.
  Arms: Free Fruit and Vegetables

SUMMARY:
The study aims to investigate whether the provision of free fresh fruits and vegetables to middle-aged men at risk of poverty increases their fruit and vegetable intake over a period of 4 weeks.

DETAILED DESCRIPTION:
A total of 100 men (> 30 years, living alone) with a low SES will be randomly assigned to a control or intervention group while controlling for food bank use. The intervention group will receive free fresh fruits and vegetables consisting of 2 daily portions of their favorite variety over a period of 4 weeks which will be provided to them once per week.

All participants will be asked to fill out a demographic questionnaire as well as a Food Frequency Questionnaire (FFQ), a questionnaire on variety of fruits and vegetables consumed and a 24-h-food-recall questionnaire. All questionnaires will be administered by trained interviewers. During the study period, the 24h-food recall questionnaire will be administered four more times; two times before the 4-week intervention period and two times after the intervention period. After the 4-week intervention period, interviewers will administered the FFQ and the questionnaire on variety.

Participants assigned to the control group will receive a fruit and vegetable basket after 4 weeks after baseline.

All participants will receive gift certificates for local supermarkets in the amount of 35,00 €.

ELIGIBILITY:
Inclusion Criteria:

* income below 980 € per month
* > 30 years of age
* living alone
* without regular food delivery service (except for e.g. meals on wheels once a day)
* born in Germany
* speaks German

Exclusion Criteria:

* lives in assisted living accommodations

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Stroebele-Benschop, PhD, Principal Investigator — Institute of Nutritional Medicine, University of Hohenheim
Locations (1):
- Institute of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Free Fruit and Vegetables: A total of four 24h-food-recall questionnaires will be administered to men (>30 years, living alone) at risk of poverty over a period of approximately 8 weeks. After baseline assessment of food intake patterns, the intervention will consist of providing free fruits and vegetables of their choice for a period of four weeks which will be provided fresh each week. At baseline and at the end of the 8-week period, a FFQ and a questionnaire on consumed fruit and vegetable amounts and variety will be administered.
  Intervention Group: The intervention consists of providing free fruits and vegetables of the participants' liking for a period of 4 weeks. Each week, a total of 2 portions of either fruits and/or vegetables per day will be provided.
- Control Goup: Control Group: A total of four 24h-food-recall questionnaires will be administered to men (>30 years, living alone) at risk of poverty over a period of approximately 8 weeks to assess their usual food intake. At baseline and at the end a 4-week period, a FFQ and a questionnaire on consumed fruit and vegetable amounts and variety will be administered.
Period: Overall Study
Arm/Group | Free Fruit and Vegetables | Control Goup
Started | 32 | 29
Completed | 25 (n=12 food bank users; n=13 non-food bank users) | 27 (n=12 food bank users; n=15 non-food bank users)
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Free Fruit and Vegetables | Control Goup | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (11.9) | 54.9 (8.5) | 54.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Variety of Fruits and Vegetables
Description: Change from Baseline in the Types of Fruit and Vegetables Consumed per Day at 4 weeks
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: types/day
Groups:
- Intervention Group: received weekly 14 portions of free fresh fruits and vegetables over a period of four weeks
- Control Group: did not receive free fresh fruits and vegetables
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 27
types/day | 2.6 (3.2) | -1.2 (3.9)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — Comparison of difference of fruit and vegetable variety between intervention group and control group

2. Primary Outcome: Amount of Fruits and Vegetables
Description: Change from Baseline in the Amount of Fruit and Vegetables Consumed per Day at 4 weeks
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: portions/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 27
portions/day | 1.1 (2.5) | -0.2 (1.3)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other; p = 0.038, Wilcoxon (Mann-Whitney) — Comparison of difference of fruit and vegetable amount between intervention group and control group

3. Secondary Outcome: Variety of Fruits and Vegetables Among Food Bank Users
Description: Change from Baseline in the Types of Fruit and Vegetables Consumed per Day at 4 weeks among food bank users.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: types/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 12
types/day | 2.2 (3.8) | -1.9 (4.6)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other; p = 0.026, Wilcoxon (Mann-Whitney) — Comparison of difference of fruit and vegetable variety between intervention group and control group

4. Secondary Outcome: Amount of Fruits and Vegetables Among Food Bank Users
Description: Change from Baseline in the Amount of Fruit and Vegetables Consumed per Day at 4 weeks among food bank users
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: portions/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 12
portions/day | 0.6 (2.2) | -0.2 (1.9)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other; p = 0.443, Wilcoxon (Mann-Whitney) — Comparison of difference of fruit and vegetable amount between intervention group and control group

5. Secondary Outcome: Variety of Fruits and Vegetables Among Non-Food Bank Users
Description: Change from Baseline in the Types of Fruit and Vegetables Consumed per Day at 4 weeks among non-Ffood Bank Users
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: types/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 15
types/day | 3.0 (2.7) | -0.7 (3.3)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other; p = 0.006, Wilcoxon (Mann-Whitney) — Comparison of difference of fruit and vegetable variety between intervention group and control group

6. Secondary Outcome: Amount of Fruits and Vegetables Among Non-Food Bank Users
Description: Change from Baseline in the Amount of Fruit and Vegetables Consumed per Day at 4 weeks among non-Food Bank Users.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: portions/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 15
portions/day | 1.5 (2.7) | -0.2 (0.8)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other; p = 0.029, Wilcoxon (Mann-Whitney) — Comparison of difference of fruit and vegetable amount between intervention group and control group

ADVERSE EVENTS:
Arm/Group | Free Fruit and Vegetables | Control Goup
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes